CLINICAL TRIAL: NCT00360152
Title: Minimally Invasive Staging of the Axilla in Breast Cancer: A Pilot Study to Assess the Feasibility of Axillary Ultrasound, Fine Needle Aspiration Biopsy and Molecular Analysis
Brief Title: Testing of Different Methods for Determining Whether Breast Cancer Has Spread to the Lymph Nodes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Society for Surgical Oncologists (Unknown); Sysmex America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-0530 / 201109077
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Axilla; Ultrasound; FNA; Molecular Analysis
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Fine-Needle; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Axillary Ultrasound (Active Comparator): Positive Axillary Ultrasound -> Fine Needle Aspiration Biopsy -> Cytopathology and Reverse Transcription-Polymerase Chain Reaction (RT-PCR) -> Positive Cyto=Axillary Lymph Node Dissection, Negative Cyto=Sentinel Lymph Node Biopsy -> Pathology
  Interventions: Procedure: Fine needle aspiration biopsy (FNAB); Procedure: Sentinel Lymph Node Biopsy
- Negative Axillary Ultrasound (Active Comparator): Negative Axillary Ultrasound -> Sentinel Lymph Node Biopsy/Fine Needle Aspiration Biopsy -> Reverse Transcription-Polymerase Chain Reaction (RT-PCR) and Pathology
  Interventions: Procedure: Fine needle aspiration biopsy (FNAB); Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Fine needle aspiration biopsy (FNAB)
Procedure: Sentinel Lymph Node Biopsy

SUMMARY:
Sentinel lymph node biopsy (SLNB) has recently emerged as a less invasive alternative to axillary lymph node dissection (ALND) in the treatment of breast cancer. However, SLNB has a number of limitations, and we believe that alternative strategies for staging of the axilla should be explored. The hypothesis of this proposal is that the combination of preoperative high-resolution axillary ultrasound (AUS), fine needle aspiration biopsy (FNAB), and molecular analysis using real-time reverse transcription-polymerase chain reaction (RT-PCR) represents a viable, minimally invasive alternative to SLNB. We propose a prospective cohort study to rigorously assess the diagnostic accuracy of molecular analysis of AUS-FNAB specimens. The primary endpoint of this study is to determine the feasibility of AUS-FNAB and real-time RT-PCR to predict the pathologic status of the axilla in a proof-of-principle study. In the short term, validation of this innovative strategy is likely to reduce the number of sentinel node procedures. In the long term, we believe that AUS-FNAB may ultimately replace SLNB.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 18 and over.
* Patients must be newly diagnosed with clinical stage I or II breast cancer and be eligible for breast surgery and core breast biopsy of their proven breast carcinoma.

Exclusion Criteria:

* Inability to give informed consent
* Contraindications for breast surgery or biopsy

Patients with no evidence of malignancy scheduled to undergo procedures under general anesthesia must fulfill the following eligibility requirements:

* Female patients, aged 18 and over
* Patient must be scheduled to undergo a procedure under general anesthesia with access to lymph nodes that can be biopsied by FNA biopsy at minimal risk to the patient
* Patient must be willing to give informed consent
* Patient with no history of malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Determine the sensitivity of AUS and real-time RT-PCR/RT-LAMP to predict the pathologic status of the axilla in breast cancer patients | At the time of ultrasound guidance and during definitive surgery for cancer
Determine the feasibility of AUS, FNAB, and RT-PCR/RT-LAMP as an alternative to SLNB for axillary staging of breast cancer patients | At the time of ultrasound guidance and during definitive surgery for cancer
Define baseline gene expression levels in lymph nodes by RT-PCR/RT-LAMP in patients with no evidence of malignancy undergoing procedures under general anesthesia | At the time of procedure under general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Margenthaler, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Valagussa P, Bonadonna G, Veronesi U. Patterns of relapse and survival following radical mastectomy. Analysis of 716 consecutive patients. Cancer. 1978 Mar;41(3):1170-8. doi: 10.1002/1097-0142(197803)41:33.0.co;2-i. PMID 638961
- [Background] Krag D, Weaver D, Ashikaga T, Moffat F, Klimberg VS, Shriver C, Feldman S, Kusminsky R, Gadd M, Kuhn J, Harlow S, Beitsch P. The sentinel node in breast cancer--a multicenter validation study. N Engl J Med. 1998 Oct 1;339(14):941-6. doi: 10.1056/NEJM199810013391401. PMID 9753708
- [Background] McMasters KM, Tuttle TM, Carlson DJ, Brown CM, Noyes RD, Glaser RL, Vennekotter DJ, Turk PS, Tate PS, Sardi A, Cerrito PB, Edwards MJ. Sentinel lymph node biopsy for breast cancer: a suitable alternative to routine axillary dissection in multi-institutional practice when optimal technique is used. J Clin Oncol. 2000 Jul;18(13):2560-6. doi: 10.1200/JCO.2000.18.13.2560. PMID 10893287
- [Background] Ung OA. Australasian experience and trials in sentinel lymph node biopsy: the RACS SNAC trial. Asian J Surg. 2004 Oct;27(4):284-90. doi: 10.1016/S1015-9584(09)60052-X. PMID 15564180
- [Background] Purushotham AD, Upponi S, Klevesath MB, Bobrow L, Millar K, Myles JP, Duffy SW. Morbidity after sentinel lymph node biopsy in primary breast cancer: results from a randomized controlled trial. J Clin Oncol. 2005 Jul 1;23(19):4312-21. doi: 10.1200/JCO.2005.03.228. PMID 15994144
- [Background] Posther KE, Wilke LG, Giuliano AE. Sentinel lymph node dissection and the current status of American trials on breast lymphatic mapping. Semin Oncol. 2004 Jun;31(3):426-36. doi: 10.1053/j.seminoncol.2004.03.019. PMID 15190501
- [Background] Fisher B, Jeong JH, Anderson S, Bryant J, Fisher ER, Wolmark N. Twenty-five-year follow-up of a randomized trial comparing radical mastectomy, total mastectomy, and total mastectomy followed by irradiation. N Engl J Med. 2002 Aug 22;347(8):567-75. doi: 10.1056/NEJMoa020128. PMID 12192016
- [Background] Brancato B, Zappa M, Bricolo D, Catarzi S, Risso G, Bonardi R, Cariaggi P, Bianchin A, Bricolo P, Rosselli Del Turco M, Cataliotti L, Bianchi S, Ciatto S. Role of ultrasound-guided fine needle cytology of axillary lymph nodes in breast carcinoma staging. Radiol Med. 2004 Oct;108(4):345-55. English, Italian. PMID 15525888
- [Background] Deurloo EE, Tanis PJ, Gilhuijs KG, Muller SH, Kroger R, Peterse JL, Rutgers EJ, Valdes Olmos R, Schultze Kool LJ. Reduction in the number of sentinel lymph node procedures by preoperative ultrasonography of the axilla in breast cancer. Eur J Cancer. 2003 May;39(8):1068-73. doi: 10.1016/s0959-8049(02)00748-7. PMID 12736105
- [Background] Krishnamurthy S, Sneige N, Bedi DG, Edieken BS, Fornage BD, Kuerer HM, Singletary SE, Hunt KK. Role of ultrasound-guided fine-needle aspiration of indeterminate and suspicious axillary lymph nodes in the initial staging of breast carcinoma. Cancer. 2002 Sep 1;95(5):982-8. doi: 10.1002/cncr.10786. PMID 12209680
- [Background] Parker SH, Dennis MA, Kaske TI. Identification of the sentinel node in patients with breast cancer. Radiol Clin North Am. 2000 Jul;38(4):809-23. doi: 10.1016/s0033-8389(05)70202-5. PMID 10943279
- [Background] Bude RO. Does contrast-enhanced US have potential for sentinel lymph node detection? Radiology. 2004 Mar;230(3):603-4. doi: 10.1148/radiol.2303031683. No abstract available. PMID 14990825
- [Background] Goldberg BB, Merton DA, Liu JB, Thakur M, Murphy GF, Needleman L, Tornes A, Forsberg F. Sentinel lymph nodes in a swine model with melanoma: contrast-enhanced lymphatic US. Radiology. 2004 Mar;230(3):727-34. doi: 10.1148/radiol.2303021440. PMID 14990839
- [Background] Wisner ER, Ferrara KW, Short RE, Ottoboni TB, Gabe JD, Patel D. Sentinel node detection using contrast-enhanced power Doppler ultrasound lymphography. Invest Radiol. 2003 Jun;38(6):358-65. PMID 12908703
- [Background] Gillanders WE, Mikhitarian K, Hebert R, Mauldin PD, Palesch Y, Walters C, Urist MM, Mann GB, Doherty G, Herrmann VM, Hill AD, Eremin O, El-Sheemy M, Orr RK, Valle AA, Henderson MA, Dewitty RL, Sugg SL, Frykberg E, Yeh K, Bell RM, Metcalf JS, Elliott BM, Brothers T, Robison J, Mitas M, Cole DJ. Molecular detection of micrometastatic breast cancer in histopathology-negative axillary lymph nodes correlates with traditional predictors of prognosis: an interim analysis of a prospective multi-institutional cohort study. Ann Surg. 2004 Jun;239(6):828-37; discussion 837-40. doi: 10.1097/01.sla.0000128687.59439.d6. PMID 15166962
- [Background] Mikhitarian K, Gillanders WE, Almeida JS, Hebert Martin R, Varela JC, Metcalf JS, Cole DJ, Mitas M. An innovative microarray strategy identities informative molecular markers for the detection of micrometastatic breast cancer. Clin Cancer Res. 2005 May 15;11(10):3697-704. doi: 10.1158/1078-0432.CCR-04-2164. PMID 15897566
- [Background] Mitas M, Mikhitarian K, Hoover L, Lockett MA, Kelley L, Hill A, Gillanders WE, Cole DJ. Prostate-Specific Ets (PSE) factor: a novel marker for detection of metastatic breast cancer in axillary lymph nodes. Br J Cancer. 2002 Mar 18;86(6):899-904. doi: 10.1038/sj.bjc.6600190. PMID 11953821
- [Background] Mitas M, Mikhitarian K, Walters C, Baron PL, Elliott BM, Brothers TE, Robison JG, Metcalf JS, Palesch YY, Zhang Z, Gillanders WE, Cole DJ. Quantitative real-time RT-PCR detection of breast cancer micrometastasis using a multigene marker panel. Int J Cancer. 2001 Jul 15;93(2):162-71. doi: 10.1002/ijc.1312. PMID 11410861
- [Background] Mitas M, Cole DJ, Hoover L, Fraig MM, Mikhitarian K, Block MI, Hoffman BJ, Hawes RH, Gillanders WE, Wallace MB. Real-time reverse transcription-PCR detects KS1/4 mRNA in mediastinal lymph nodes from patients with non-small cell lung cancer. Clin Chem. 2003 Feb;49(2):312-5. doi: 10.1373/49.2.312. No abstract available. PMID 12560358
- [Background] Wallace MB, Block MI, Gillanders W, Ravenel J, Hoffman BJ, Reed CE, Fraig M, Cole D, Mitas M. Accurate molecular detection of non-small cell lung cancer metastases in mediastinal lymph nodes sampled by endoscopic ultrasound-guided needle aspiration. Chest. 2005 Feb;127(2):430-7. doi: 10.1378/chest.127.2.430. PMID 15705978
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu